CLINICAL TRIAL: NCT00631644
Title: Eating Behavior in Adolescents
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080085; 08-CH-0085
Record Dates: First submitted 2008-03-07; First posted 2008-03-10 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2015-09-08

CONDITIONS: Overweight; Eating Behavior; Binge Eating
Keywords: Adolescents; Eating Behavior; Eating in the Absence of Hunger; Disordered Eating; Food Intake; Macronutrient Composition; Obesity; Adolescent; Healthy Volunteer; HV
MeSH Terms: conditions — Overweight; Feeding Behavior; Bulimia; Obesity

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will explore the eating habits of adolescents and determine if eating behavior is linked to genetics.

Healthy adolescents between 13 and 17 years of age may be eligible for this study. Candidates come to the NIH Clinical Center at 8:00 AM to be screened with the following:

* Medical history and brief physical examination, including height, weight, and body fat measurements. Body fat is measured using a device called a Bod Pod. The adolescent sits inside the device for about 5 minutes and the machine determines body fat by measuring air movement. The adolescent must wear a tight-fitting swimsuit for this test.
* Urine test to look for sugar or protein in the urine and to test for pregnancy in females.
* Blood tests for routine chemistries and for gene studies related to eating behaviors.
* Questionnaires and interviews about the adolescent s general health and eating habits.
* Acclimatization to test meal conditions for the study. The adolescent is given a breakfast shake to drink.

Participants come to the NIH Clinical Center at 10:30 AM for laboratory meal testing. At this visit, the adolescent does the following:

* Eats food from a buffet of everyday foods that most kids eat.
* Fills out questionnaires.
* Tastes and rates the flavor of a variety of snack foods.

DETAILED DESCRIPTION:
Little is known about the eating behaviors that place adolescents at heightened risk for overweight. In the proposed study, we aim to investigate the role that eating behaviors and genes may play in the development of overweight. Participants will be adolescent girls and boys from a racially/ethnically diverse sample of adolescents from the DC Metro community. Adolescent eating behavior will be observed during laboratory test meals. Adolescents will be provided with a large buffet of foods or a standard meal and instructed to eat until you are no longer hungry. Thirty minutes later, they will taste and rate a variety of highly palatable snack foods. Blood tests will be conducted to examine genes related to eating behavior. Assessments also will include affective states, degree of hunger, degree of fullness, body image satisfaction, disordered eating attitudes and behaviors, and measures of interpersonal interactions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify for participation in the study if they meet the following criteria:

1. <TAB>Age 13-17 years.
2. <TAB>Good general health as indicated by medical history and physical examination.
3. <TAB>Negative urine glucose and normal electrolytes, hepatic, and thyroid function.
4. <TAB>For the fMRI portion only: right handedness (required for standardization of responses).
5. <TAB>For the fMRI portion only: female.
6. <TAB>For the fMRI portion only: overweight (BMI greater than or equal to 85th percentile for age and sex).

EXCLUSION CRITERIA:

Volunteers will be excluded if they have any of the following:

1. <TAB>Medical problem likely to affect caloric intake.
2. <TAB>History of any condition including psychiatric disorders in either child or their responsible parent that in the opinion of the investigators would impede competence to sign consent, interfere with adherence to procedures, or possibly hinder completion of the study.
3. <TAB>Pregnancy.
4. <TAB>Use of medication likely to affect caloric intake.
5. <TAB>History of significant neurological injury or insult.
6. <TAB>For the fMRI portion only: braces (or other metal) that would interfere with the fMRI procedure.
7. <TAB>For the fMRI portion only: non-native English speakers (required for standardization of responses).

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2008-03-05; Study Completion 2015-09-08

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Barros A. [Individual impression spoon from self polymerising plastics]. Zahnarztl Prax. 1967 Jan 1;18(1):1. No abstract available. German. PMID 5340113
- [Background] Taylor ED, Theim KR, Mirch MC, Ghorbani S, Tanofsky-Kraff M, Adler-Wailes DC, Brady S, Reynolds JC, Calis KA, Yanovski JA. Orthopedic complications of overweight in children and adolescents. Pediatrics. 2006 Jun;117(6):2167-74. doi: 10.1542/peds.2005-1832. PMID 16740861
- [Derived] Suelter CS, Schvey N, Kelly NR, Shanks M, Thompson KA, Mehari R, Brady S, Yanovski SZ, Melby CL, Tanofsky-Kraff M, Yanovski JA, Shomaker LB. Relationship of pressure to be thin with gains in body weight and fat mass in adolescents. Pediatr Obes. 2018 Jan;13(1):14-22. doi: 10.1111/ijpo.12179. Epub 2016 Nov 16. PMID 27860465
- [Derived] Schvey NA, Shomaker LB, Kelly NR, Pickworth CK, Cassidy O, Galescu O, Demidowich AP, Brady SM, Tanofsky-Kraff M, Yanovski JA. Pressure To Be Thin and Insulin Sensitivity Among Adolescents. J Adolesc Health. 2016 Jan;58(1):104-10. doi: 10.1016/j.jadohealth.2015.09.010. PMID 26707232
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388
- [Derived] Vannucci A, Tanofsky-Kraff M, Ranzenhofer LM, Kelly NR, Hannallah LM, Pickworth CK, Grygorenko MV, Brady SM, Condarco TA, Kozlosky M, Demidowich AP, Yanovski SZ, Shomaker LB, Yanovski JA. Puberty and the manifestations of loss of control eating in children and adolescents. Int J Eat Disord. 2014 Nov;47(7):738-47. doi: 10.1002/eat.22305. Epub 2014 May 30. PMID 24888295
- [Derived] Reina SA, Shomaker LB, Mooreville M, Courville AB, Brady SM, Olsen C, Yanovski SZ, Tanofsky-Kraff M, Yanovski JA. Sociocultural pressures and adolescent eating in the absence of hunger. Body Image. 2013 Mar;10(2):182-90. doi: 10.1016/j.bodyim.2012.12.004. Epub 2013 Feb 7. PMID 23394966
- [Derived] Shomaker LB, Tanofsky-Kraff M, Zocca JM, Courville A, Kozlosky M, Columbo KM, Wolkoff LE, Brady SM, Crocker MK, Ali AH, Yanovski SZ, Yanovski JA. Eating in the absence of hunger in adolescents: intake after a large-array meal compared with that after a standardized meal. Am J Clin Nutr. 2010 Oct;92(4):697-703. doi: 10.3945/ajcn.2010.29812. Epub 2010 Aug 18. PMID 20720255